CLINICAL TRIAL: NCT00377819
Title: A Randomized Study to Evaluate Safety and Efficacy of Transitioning Therapy From Alendronate to Denosumab (AMG 162) in Postmenopausal Women With Low Bone Mineral Density
Brief Title: Study of Transitioning From Alendronate to Denosumab
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20050234
Record Dates: First submitted 2006-09-14; First posted 2006-09-18 (Estimated); Results first posted 2010-08-03 (Estimated); Last update posted 2011-07-11 (Estimated); Status verified 2011-06

CONDITIONS: Postmenopausal Osteoporosis
Keywords: RANKL; RANK; denosumab; AMG 162; osteoporosis; bone turnover; bone mineral density; clinical trial; postmenopausal osteoporosis; alendronate; total hip bone mineral density
MeSH Terms: conditions — Osteoporosis, Postmenopausal; Osteoporosis | interventions — Alendronate; Denosumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- denosumab (Experimental)
  Interventions: Drug: Denosumab (AMG 162)
- alendronate (Active Comparator)
  Interventions: Drug: alendronate

INTERVENTIONS:
Drug: alendronate — 70 mg oral QW
  Arms: alendronate
Drug: Denosumab (AMG 162) — 60 mg SC q 6 mos
  Arms: denosumab

SUMMARY:
The study will evaluate the efficacy and safety of transitioning postmenopausal women on current alendronate therapy to denosumab. Endpoints studied will include bone mineral density, bone turnover markers and bone histology in a subset of subjects.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal females 55 yrs or older
* Received alendronate therapy for osteoporosis for at least 6 months prior to entry into study
* Lumbar spine or total hip Bone Mineral Density (BMD) corresponding to T-score ≤ -2 and ≥ -4

Exclusion Criteria:

* Vitamin D deficiency
* Administration of intravenous bisphosphonate, or
* fluoride (except for dental treatment) or
* strontium ranelate
* Administration of Parathyroid Hormone (PTH) or Parathyroid Hormone (PTH) derivatives (eg; teriparatide) within the last year
* Administration of any bisphosphonate other than alendronate (ALN) within 1 year of screening

Min Age: 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 504 (Actual)
Dates: Start 2006-09; Primary Completion 2008-03 (Actual); Study Completion 2008-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- [Result] Kendler DL, Roux C, Benhamou CL, Brown JP, Lillestol M, Siddhanti S, Man HS, San Martin J, Bone HG. Effects of denosumab on bone mineral density and bone turnover in postmenopausal women transitioning from alendronate therapy. J Bone Miner Res. 2010 Jan;25(1):72-81. doi: 10.1359/jbmr.090716. PMID 19594293
- [Derived] Miller PD, Pannacciulli N, Malouf-Sierra J, Singer A, Czerwinski E, Bone HG, Wang C, Huang S, Chines A, Lems W, Brown JP. Efficacy and safety of denosumab vs. bisphosphonates in postmenopausal women previously treated with oral bisphosphonates. Osteoporos Int. 2020 Jan;31(1):181-191. doi: 10.1007/s00198-019-05233-x. Epub 2019 Nov 28. PMID 31776637
- [Derived] Gold DT, Horne R, Coon CD, Price MA, Borenstein J, Varon SF, Satram-Hoang S, Macarios D. Development, reliability, and validity of a new Preference and Satisfaction Questionnaire. Value Health. 2011 Dec;14(8):1109-16. doi: 10.1016/j.jval.2011.06.010. Epub 2011 Oct 1. PMID 22152181
- [Derived] Reid IR, Miller PD, Brown JP, Kendler DL, Fahrleitner-Pammer A, Valter I, Maasalu K, Bolognese MA, Woodson G, Bone H, Ding B, Wagman RB, San Martin J, Ominsky MS, Dempster DW; Denosumab Phase 3 Bone Histology Study Group. Effects of denosumab on bone histomorphometry: the FREEDOM and STAND studies. J Bone Miner Res. 2010 Oct;25(10):2256-65. doi: 10.1002/jbmr.149. PMID 20533525
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First Subject Enrolled: 02-Oct-2006 Last Subject Enrolled: 07-Mar-2007
Groups:
- Alendronate 70 mg QW: 70 mg alendronate once weekly (QW) orally plus placebo for denosumab subcutaneously once every 6 months (Q6M)
- Denosumab 60 mg Q6M: 60 mg denosumab administered subcutaneously once every 6 months (Q6M) plus placebo for alendronate once weekly (QW) orally
Period: Overall Study
Arm/Group | Alendronate 70 mg QW | Denosumab 60 mg Q6M
Started | 251 | 253
Received Study Medication | 249 | 253
Completed | 238 | 243
Not Completed | 13 | 10
Not completed — Adverse Event | 2 | 3
Not completed — Withdrawal by Subject | 10 | 4
Not completed — Death | 0 | 1
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Alendronate 70 mg QW | Denosumab 60 mg Q6M | Total
Number analyzed (Participants) | 251 | 253 | 504
Age Continuous [Mean (Standard Deviation); unit: Years] | 68.2 (7.7) | 66.9 (7.8) | 67.6 (7.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 251 | 253 | 504
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants]
  White or Caucasian | 232 | 238 | 470
  Black or African American | 2 | 0 | 2
  Hispanic or Latino | 12 | 11 | 23
  Asian | 1 | 1 | 2
  Japanese | 1 | 3 | 4
  American Indian or Alaska Native | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Other | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Total Hip Bone Mineral Density
Description: Bone Mineral Density Assessed by Dual Energy X-Ray Absorptiometry. Percent change calculated using [(12 month value - baseline value) / baseline value]*100.
Time Frame: Baseline, 12 months
Population: Participants with non-missing baseline evaluation and at least 1 non-missing post-baseline evaluation.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Alendronate 70 mg QW | Denosumab 60 mg Q6M
Number analyzed (Participants) | 233 | 241
Percent Change | 1.05 [0.76 to 1.34] | 1.9 [1.61 to 2.18]
Statistical Analysis 1: Comparison: Alendronate 70 mg QW vs Denosumab 60 mg Q6M; Test type: Non-Inferiority or Equivalence — Non-inferiority margin = -0.35%; p < 0.0001, Repeated Measures Model; Mean Difference (Final Values) = 0.85, 95% CI [0.44 to 1.25] — Based on repeated measures model adjusting for treatment, length of prior alendronate stratification variable, visit, baseline value, machine type, treatment by visit interaction, and baseline value by machine type interaction

2. Secondary Outcome: Percent Change From Baseline in Lumbar Spine Bone Mineral Density
Description: as for outcome 1
Time Frame: Baseline, 12 months
Population: Participants with non-missing baseline evaluation and at least 1 non-missing post-baseline evaluation.
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent Change
Arm/Group | Alendronate 70 mg QW | Denosumab 60 mg Q6M
Number analyzed (Participants) | 235 | 242
Percent Change | 1.85 [1.44 to 2.26] | 3.03 [2.63 to 3.44]
Statistical Analysis 1: Comparison: Alendronate 70 mg QW vs Denosumab 60 mg Q6M; Test type: Non-Inferiority or Equivalence — Non-inferiority margin = -0.22%; p < 0.0001, Repeated Measures Model; Mean Difference (Final Values) = 1.18, 95% CI [0.63 to 1.73] — [estimate comment as in outcome 1, analysis 1]

3. Secondary Outcome: Percent Change From Baseline in Serum C-Telopeptide-I (CTX-I)
Description: Percent Change From Baseline to Month 3 in Serum CTX-I. Percent change calculated using [(3 month value - baseline value) / baseline value]*100.
Time Frame: Baseline, 3 months
Population: Participants with non-missing baseline evaluation and non-missing post-baseline evaluation at month 3.
Measure: Median (Inter-Quartile Range); unit: Percent Change
Arm/Group | Alendronate 70 mg QW | Denosumab 60 mg Q6M
Number analyzed (Participants) | 240 | 245
Percent Change | -4.2 [-29.4 to 25.1] | -63.3 [-78.5 to -38.0]
Statistical Analysis 1: Comparison: Alendronate 70 mg QW vs Denosumab 60 mg Q6M; Test type: Superiority or Other; p < 0.0001, Van Elteren Stratified Rank Test

ADVERSE EVENTS:
Time Frame: 12 months
Description: The table of Other Adverse Events summarizes the most frequent non-serious occurrences of adverse events.
Arm/Group | Alendronate 70 mg QW | Denosumab 60 mg Q6M
Serious Adverse Events (participants affected / at risk) | 16/249 | 15/253
Other Adverse Events (participants affected / at risk) | 101/249 | 103/253
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Alendronate 70 mg QW (N=249) | Denosumab 60 mg Q6M (N=253)
Angina pectoris (Cardiac disorders) | 1 | 1
Atrial fibrillation (Cardiac disorders) | 1 | 0
Atrial flutter (Cardiac disorders) | 0 | 1
Sick sinus syndrome (Cardiac disorders) | 0 | 1
Appendicitis perforated (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Loose tooth (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
Hyperpyrexia (General disorders) | 1 | 0
Inflammation (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1
Anaphylactic reaction (Immune system disorders) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Diverticulitis (Infections and infestations) | 0 | 1
Gingival infection (Infections and infestations) | 1 | 0
Lobar pneumonia (Infections and infestations) | 1 | 0
Periodontal infection (Infections and infestations) | 1 | 0
Foot fracture (Injury, poisoning and procedural complications) | 0 | 1
Head injury (Injury, poisoning and procedural complications) | 1 | 0
Tooth fracture (Injury, poisoning and procedural complications) | 2 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 1
Synovitis (Musculoskeletal and connective tissue disorders) | 0 | 1
Ameloblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Nodular fasciitis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Carotid artery stenosis (Nervous system disorders) | 0 | 1
Cerebrovascular accident (Nervous system disorders) | 1 | 1
Cystocele (Reproductive system and breast disorders) | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | 1 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Hypertension (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Alendronate 70 mg QW (N=249) | Denosumab 60 mg Q6M (N=253)
Constipation (Gastrointestinal disorders) | 12 | 13
Bronchitis (Infections and infestations) | 14 | 16
Nasopharyngitis (Infections and infestations) | 27 | 34
Arthralgia (Musculoskeletal and connective tissue disorders) | 26 | 15
Back pain (Musculoskeletal and connective tissue disorders) | 29 | 27
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 13 | 11
Pain in extremity (Musculoskeletal and connective tissue disorders) | 21 | 12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Clinical Trial Agreement generally does not restrict an investigator's discussion of trial results after completion. The Agreement permits Amgen a limited period of time to review material discussing trial results (typically up to 45 days and possible extension). Amgen may remove confidential information, but authors have final control and approval of publication content. For multi-center studies, the investigator agrees not to publish any results before the first multi-center publication.